CLINICAL TRIAL: NCT02780856
Title: Clinical Study to Evaluate the Safety and Performance of the Calcivis System for Identifying Active Demineralization on Tooth Surfaces
Brief Title: Safety and Performance Evaluation of the Calcivis System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calcivis Ltd (Industry)
Collaborators: Medsource UK Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAL-02-2014
Record Dates: First submitted 2016-05-12; First posted 2016-05-24 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Dental Caries
Keywords: Caries Activity Demineralisation; Demineralisation
MeSH Terms: conditions — Dental Caries | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sound and unsound teeth (Other): Sound (ICDAS 0) canines or incisors and unsound (ICDAS 2 or 3) molars or pre-molars - imaging with the Calcivis System
  Interventions: Device: Imaging with the Calcivis System

INTERVENTIONS:
Device: Imaging with the Calcivis System — Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried and a black & white and luminescent image of each tooth taken. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
  Other Names: Calcivis Caries Activity Imaging System

SUMMARY:
This is a prospective, multi-centre clinical study to evaluate the safety and performance of the Calcivis Caries Activity Imaging System. Dentists will identify tooth surfaces as either sound (inactive) or unsound (active caries lesion present) according to ICDAS staging (International Caries Detection and Assessment System). Images of the tooth surface will be taken with the Calcivis System immediately before and after application of a disclosing solution containing a bioluminescent protein. Presence or absence of elevated luminescence on the images will indicate activity / inactivity of the presence or absence of active demineralisation on the tooth surfaces.

The study will be deemed a success if there is 70% agreement and above between:

1. elevated luminescence and the presence of active caries as determined by the dentists, and
2. absence of luminescence and the determination of a sound tooth surface by the dentists.

DETAILED DESCRIPTION:
Dental caries (tooth decay) is a significant clinical and public health problem. The development of caries lesions involves a net mineral loss of dental tissue, which can lead to progressive loss of tooth structure and associated pain and disease. Detecting, assessing, diagnosis and treating such lesions are core activities in dentistry. Currently the main detection and diagnosis aids are visual inspection and the used of a probe, together with X-ray images. Determination of the activity status of a lesion (how likely it is to progress) is required to assess treatment needs. Currently methods are problematic and involve the clinicians' subjective assessment and / or monitoring of lesions progression over a number of visits.

A previous clinical study on the prototype of the Calcivis System has been conducted. The results concluded that the Calcivis System was safe for use and the level of agreement between elevated luminescence and areas of expected activity was above 70% and not due to chance (NCT02098304).

This prospective, multi-centre clinical study has been designed to assess the safety and performance of the Calcivis System. The device under evaluation comprises a hand-held customized intra-oral camera which takes images of a lesion on a tooth surface immediately before and after application of a disclosing solution which contains a bioluminescent photo-protein. The photo-protein detects free calcium ions on the tooth surface and produces a light signal if the caries lesion is active.

For the clinical study, patients identified by the Investigator from those attending routine dental appointments, who meet all the inclusion and exclusion criteria will be approached to discuss their possible participation in the study. Patients will be given a Patient Information Sheet to read and time to consider their participation in the study. If they are happy to participate they will attend for two Study Visits, 7 to 14 days apart. Written informed consent will be taken before any study procedures are conducted. As children under the age of 16 are included in this study, parent / guardian consent will be taken where appropriate.

At study Visit 1, demographics, relevant medications and oral hygiene data will be collected. The dentist will carry out an oral examination and the tooth / teeth identified as per inclusion / exclusion criteria, will be cleaned with prophy paste, rinsed with tap water and a 3-in-1 air / water spray before being air dried and staged as per ICDAS coding. Reference intra-oral photographs will be taken of each tooth. The tooth / teeth surfaces will again be air dried before imaging with the Calcivis System, immediately before and after application of the disclosing solution. A maximum of one sound (unrestored, accessible, free smooth surface of a canine or incisor, away from the gingival margin with no visible caries lesion) and one unsound (erupting or erupted molar or premolar with a visible lesion deemed to be active, in a plaque stagnation area) tooth will be imaged per patient. after imaging is completed, patients rinse out with tap water. Adverse events will be collected throughout. The dentist will then share the Calcivis images of the teeth with the patient. Post imaging questionnaires will be completed by each patient at the end of Study Visit 1 and user questionnaires completed by the dental team at the end of each Study Visit 1 day.

Patients will return for (Study Visit 2), 7 to 14 days after Visit 1, when a final oral examination will take place. Any adverse events observed or volunteered by the patient will be recorded.

The study images will be independently reviewed by another dentist, for agreement between expected lesion activity / inactive teeth and the Calcivis System.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 6 years or older
2. Patient must have one unrestored, accessible, free smooth buccal surface on a canine or incisor, away from the gingival surface identified with no visible lesions (coded ICDAS 0) and/or
3. Patient must have one unrestored, accessible, erupting or erupted molar or premolar with a visible lesion identified as (coded ICDAS 2 or 3) in a plaque stagnation area
4. Patient and / or parent or guardian must be willing and able to give written informed consent
5. Patient and / or parent or guardian must be willing and able to adhere to study schedule

Exclusion Criteria:

1. Any patient with recent tooth bleaching (within previous two weeks of imaging with the Calcivis System)
2. Any patient having on-going re-mineralization treatment including, but not limited to high concentration prescription fluoride toothpaste
3. Any patient with a fixed orthodontic appliance
4. Any patient currently taking part in a clinical research study, or has taken part in a clinical research study in the previous three months
5. Pregnant and / or nursing mothers

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-01-14 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Shanks, BDS, MJDF, Study Director — Harper, Downie and Shanks Dental Practice; Elaine Downie, BDS, Principal Investigator — Harper, Downie and Shanks Dental Practice; Fraser Morrison, BDS, Principal Investigator — Bathgate Smile Centre; Steve Martin, BDS, MJDF, Principal Investigator — Edinburgh Periodontics; Agnieszka Nohawica, BDS, Principal Investigator — Bosco Dental Studio
Locations (4):
- United Kingdom (4):
  - Bosco Dental Studio, Dalkeith, Edinburgh
  - Bathgate Smile Centre, Bathgate
  - Harper, Downie and Shanks Dental Practice, Edinburgh
  - Edinburgh Periodontics, Edinburgh

IPD SHARING:
Plan to Share IPD: No
A Final Clinical Study report will be issued

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by 5 Investigators from 4 UK, dental practices between 14 January and 04 May 2017.
  110 patients attended Visit 1 and were imaged with the Calcivis System, therefore data from 110 patients are included in the safety and agreement populations.
Units Other Than Participants: Teeth
Groups:
- Sound and Unsound Teeth: Sound (ICDAS 0) canines or incisors and unsound (ICDAS 2 or 3) molars or pre-molars - imaging with the Calcivis System
  Imaging with the Calcivis System: Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried. Both black & white and luminescent images will be taken. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Period: Overall Study
Arm/Group | Sound and Unsound Teeth
Started (Attended Visit 1 when teeth were imaged with the Calcivis System) | 110; 176 Teeth
Completed (Attended Visit 2 - no images taken at this visit) | 109; 176 Teeth
Not Completed | 1; 0 Teeth
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients six years or older were recruited who had one unrestored, accessible free smooth buccal surface on a canine or incisor away from gingival surface identified with no lesion (ICDAS 0) and / or one unrestored, accessible, erupting or erupted molar or pre-molar with a visible lesion (ICDAS 2 or 3) in a plaque stagnation area
Units Other Than Participants: Teeth
Groups:
- Sound and Unsound Teeth: Sound (ICDAS 0) canines or incisors and unsound (ICDAS 2 or 3) molars or pre-molars - imaging with the Calcivis System
  Imaging with the Calcivis System: Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried and both black & white and luminescent images of each tooth taken.The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Sound and Unsound Teeth
Number analyzed (Participants) | 110
Number analyzed (Teeth) | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Asian | 2
  Black | 1
  White | 107
  Other | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 110
Sound (inactive)and unsound (active) teeth [Count of Units; unit: Teeth]
  Number of sound teeth | 90
  Number of unsound teeth | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Teeth Identified as Sound or Unsound by the Calcivis System That Were in Agreement With the Dentist's Assessment
Description: Agreement between the dentist's assessment (ICDAS staging) of sound (inactive) and unsound (active) teeth and the visible presence of elevated bioluminescence on the tooth surface using the Calcivis System
Time Frame: Day 0
Population: From the 110 patients recruited and imaged with the Calcivis System, 90 provided a sound tooth (ICDAS 0) and 86 provided an unsound tooth (ICDAS 2 or 3) with interpretable images were included in the Primary Agreement Analysis
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Groups:
- Sound: Sound (ICDAS 0) canines or incisors - imaging with the Calcivis System
  Imaging with the Calcivis System: Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried and both black & white and luminescent images taken. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
- Unsound: Unsound (ICDAS 2 or 3) molars or premolars - imaging with the Calcivis System
  Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried and both black & white and luminescent images taken. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Sound | Unsound
Number analyzed (Participants) | 90 | 86
Number analyzed (teeth) | 90 | 86
teeth | 88 | 78
Statistical Analysis 1: Comparison: Sound; The null and alternative hypothesis for each tooth population was of chance agreement (50%) and was tested against an exact binomial one-sided 97.5% confidence interval; Test type: Superiority; p < 0.0001, exact binomial; An exact binomial test was used and an exact 97.5% Confidence Level using the Clopper-Pearson method was calculated
Statistical Analysis 2: Comparison: Unsound; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, exact binomial; An exact binomial test was used and an exact 97.5% Confidence Level using the Clopper-Pearson method was calculated

2. Primary Outcome: Number of Non-patient Related Adverse Events of the Calcivis System
Description: Collection of all Adverse Events throughout the duration of the study
Time Frame: Day 0 and Day 7
Population: All patients on whom the Calcivis System has been used
Measure: Number; unit: adverse events
Groups:
- Sound and Unsound Teeth: Sound (ICDAS 0) canines or incisors and unsound (ICDAS 2 or 3) molars or pre-molars - imaging with the Calcivis System
  Imaging with the Calcivis System: Following identification of both sound and unsound teeth, both black & white and luminescent images were taken. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Sound and Unsound Teeth
Number analyzed (Participants) | 110
adverse events | 3

3. Secondary Outcome: Patient Experience
Description: Completion of Patient Questionnaires after imaging with the Calcivis System
Time Frame: Day 0
Population: Patient Questionnaires were completed for all 110 patients imaged at Visit 1 and comprised two questions and the patient was asked to tick the most appropriate response on a three-point scale e.g. good, neither good nor bad, bad etc
Measure: Count of Units; unit: patient questionnaires
Units Other Than Participants: patient questionnaires
Groups:
- Sound and Unsound Teeth: Imaging of sound (ICDAS 0) canines or incisors and unsound (ICDAS 2 or 3) molars or pre-molars with the Calcivis System
  Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried and both black & white and luminescent images taken. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Sound and Unsound Teeth
Number analyzed (Participants) | 110
Number analyzed (patient questionnaires) | 110
patient questionnaires
  Calcivis System experience: good | 93
  Calcivis System experience:neither good nor bad | 17
  Calcivis System experience:bad | 0
  Image review with Dentist: helpful | 106
  ImagereviewwithDentist:neitherhelpfulnorunhelpful | 4
  Image review with Dentist:unhelpful | 0

4. Secondary Outcome: User Experience
Description: Completion of User Questionnaires after imaging with the Calcivis system
Time Frame: Day 0
Population: User Questionnaires were completed by the dentist and nurse at the end of every imaging session about their experiences using the Calcivis System. Imaging sessions could include one or several participants, therefore multiple participants could be accounted for in a single User Questionnaire providing 61 questionnaires covering 110 participants.
Measure: Count of Units; unit: User Questionnaires
Units Other Than Participants: User Questionnaires
Arm/Group | Sound and Unsound Teeth
Number analyzed (Participants) | 110
Number analyzed (User Questionnaires) | 61
User Questionnaires
  Calcivis System preparation:easy | 49
  CalcivisSystempreparation:neithereasynordifficult | 9
  Calcivis System preparation: difficult | 3
  Calcivis System use:easy | 34
  Calcivis System use: neither easy nor difficult | 19
  Calcivis System use: difficult | 8
  Calcivis System experience: good | 30
  Calcivis System experience: neither good nor bad | 25
  Calcivis System experience: bad | 6
  Ease of use of IFU: easy | 52
  Ease of use of IFU: neither easy nor difficult | 9
  Ease of use of IFU: difficult | 0

ADVERSE EVENTS:
Time Frame: 7 to 14 days
Description: All adverse events and device deficiencies were collected throughout the study on Adverse Event Forms
Groups:
- Sound and Unsound Teeth: Sound (ICDAS 0) canines or incisors and unsound (ICDAS 2 or 3) molars or pre-molars - imaging with the Calcivis System
  Imaging with the Calcivis System: Following identification of both sound and unsound tooth surfaces, the teeth will be air-dried and images of each tooth taken immediately before and after application of a small amount of disclosing solution. The images of each tooth will be overlaid and a resulting demineralization map of the tooth produced, indicating areas of elevated bioluminescence corresponding to free calcium ions on the surface of the tooth (active caries)
Arm/Group | Sound and Unsound Teeth
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 3/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sound and Unsound Teeth (N=110)
Device Deficiency (Product Issues) | 3 (3) — Device Deficiency - inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT02780856/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02780856/SAP_001.pdf